CLINICAL TRIAL: NCT04788134
Title: Normative Data for Post-rotatory Nystagmus Test at Spanish Adolescent and Adult Population: a Transversal Study
Brief Title: Post- Rotatory Nystagmus Test: Normative Data for Spanish Adolescents and Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Quesada, Rocío Vico (Individual)
Responsible Party: Principal Investigator, Rocío Vico Quesada, Quesada, Rocío Vico, Quesada, Rocío Vico
Other Study IDs: 010395
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Vestibular Function Tests; Nystagmus Vestibular
Keywords: vestibular function tests; nystagmus, physiologic; adult; adolescent
MeSH Terms: conditions — Nystagmus, Pathologic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Post-rotatory nystagmus test — The test is administrated with the person sit down with cross legs at a rotatory board, with the head positioned by the examiner in 30° of forward flexion. The position was maintained by the administration of the test. The administration consist in two administrations separate by one minute. Each administration consist in rotate the person 10 times in 20 seconds (the first 10 rotations in a counterclockwise direction in 20 s and the second 10 rotations in a clockwise direction in 20 s). After each administration the examiner counts the duration of the reflex in seconds.

SUMMARY:
The vestibulo-ocular reflex is the motor response of our eyes in the opposite direction to a translational or rotational movement of our head. The post-rotational nystagmus test (PRN) assesses the integrity of this reflex, thus assessing the perception of the vestibular system. The duration of this reflex after administering this test has been widely studied in children from 2 months to 12 years and 11 months of age. However, there is a knowledge gap from that age that the present study seeks to address.

DETAILED DESCRIPTION:
The vestibulo-ocular reflex (VOR) is the motor response of our eyes in the opposite direction to a translational or rotational movement of our head. The post-rotational nystagmus test (PRN) assesses the integrity of this reflex, thus assessing the perception of the vestibular system. This system has an important role in our balance, stabilization of the visual field when our head moves, awareness of the position of our head in space, postural control and functions of the Autonomous Nervous System.

The duration of this reflex after administering this test has been widely studied in children from 2 months to 12 years and 11 months of age. However, there is a knowledge gap from that age that the present study seeks to address. This article aims to explore the use of the PRN test for adolescent and adults, to prove if the duration of the VOR is longer in these population than in children. It will be also recollected personal data to study whether exposure to vestibular input influences its reactivity and perception.

ELIGIBILITY:
Inclusion Criteria:

* People over 13 years of age.
* Spanish-speaking population.
* Signature of the informed consent.

Exclusion Criteria:

* Diagnosis of a neurodevelopmental or neurological disorder.
* Being in occupational therapeutic treatment for balance or vestibular problems.
* Practice of sports in one previous hour.
* Adverse reaction to vestibular input such as vomiting, discoloration, feeling of unpleasantness or any other type of negative reaction before / during / after the administration of the NPR.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People over 13 years, that lives in the north, middle and south of Spain, and meet the selection criteria.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Duration of vestibular-ocular reflex after the administration of nystagmus post-rotatory test in adolescent and adult population | End of the nystagmus post rotatory test and end of the vestibular-ocular reflex
  The post rotatory nystagmus test evaluates the duration of the vestibular-ocular reflex: how long its lats gives information about the perception of vestibular system. This reflex reflects the role of the vestibular system in ocular mechanisms (Mailloux et al., 2014). It is administered twice: clockwise and counterclockwise.After the administration the physiologic nystagmus appears, it is our vestibular-ocular reflex, and the examiner has to register the duration of it.

CONTACTS AND LOCATIONS:
Overall Officials: Vico Rocío, Principal Investigator — Quesada, Rocío Vico; Pedrero Yolanda, Principal Investigator — Quesada, Rocío Vico; Zisa Nerina, Principal Investigator — Quesada, Rocío Vico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mailloux Z, Leao M, Becerra TA, Mori AB, Soechting E, Roley SS, Buss N, Cermak SA. Modification of the postrotary nystagmus test for evaluating young children. Am J Occup Ther. 2014 Sep-Oct;68(5):514-21. doi: 10.5014/ajot.2014.011031. PMID 25184463